CLINICAL TRIAL: NCT06581835
Title: Accuracy Performance Verification of the INVOS™ PM7100 System by Comparing rSO2 Values to Reference Blood Oxygen Saturation Measurements in Adult Human Volunteers
Brief Title: Accuracy Performance Verification of the INVOS™ PM7100 System in Adults
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT23038INSENS
Record Dates: First submitted 2024-08-23; First posted 2024-09-03 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2024-07

CONDITIONS: Oxygen Saturation
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Observational: Healthy, non-smoking volunteers ages 18-50 years who meet inclusion criteria
  Interventions: Device: Observational

INTERVENTIONS:
Device: Observational — The study objective requires placement of a jugular venous bulb catheter in the right or left jugular venous bulb with ultrasound guidance. A venous and radial arterial line will be placed. Two INVOS™ sensors (PMSENS71-A) will be placed bilaterally on the subject's forehead. The INVOS™ device will be evaluated for a targeted range of 70-100% SpO2 levels. Hypoxic mixtures of gas are delivered, and data are collected at approximately (~) 5-minute intervals during steady periods of increasing and decreasing oxygen concentration.

SUMMARY:
Prospective, observational, post-market, verification study to ensure compliance to the ISO 80601-2-85:2021 standard

DETAILED DESCRIPTION:
The purpose of this study is to provide data for verification of the INVOS™ PM7100 System paired with the Adult Sensor (PMSENS71-A). Medtronic evaluates the performance and/or feasibility of non-invasive optical devices over a clinically relevant range of arterial saturations. This study evaluates rSO2 accuracy of tissue oximetry equipment compared directly to the actual saturation of arterial and jugular blood samples (SaO2) and (SjvO2) and the composite of the two (SavO2) as measured by co-oximetry.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 18 to 50 years
2. Completion of a health screening for medical history by a licensed physician, nurse practitioner, or physician assistant
3. Minimum weight 40kg
4. BMI within range 18.0 - 29.9

Exclusion Criteria:

1. Prior or known allergies to lidocaine (or similar pharmacologic agents, e.g., Novocain) [self-reported]
2. Prior known severe allergies to medical grade adhesive/tape (Band-Aid) [self-reported]
3. Subjects taking medication(s) beyond birth control may be excluded from participating at the PI discretion [self-reported]
4. Any interventional study within 30 days that, in the opinion of the PI, electrocardiogram (ECG) may interfere with study participation (i.e., drug, biologic)
5. Negative Allen's test for radial and ulnar patency
6. Has made a whole blood donation or has had at least 450 ml of blood drawn within 8 weeks prior to the study procedure [self-reported]
7. Is pregnant
8. Has anemia as measured by co-oximetry [values specific for sex]
9. Has a history of sickle cell trait or thalassemia [self-reported]
10. Has an abnormal hemoglobin electrophoresis test [lab measurement]
11. Has a positive urine cotinine test or urine drug screen or oral ethanol test [Point of Care (POC) testing]
12. Has a room air saturation less than 95% by pulse oximetry [measurement by PI or delegate]
13. Has a clinically significant abnormal ECG [assessment by PI or delegate]
14. Has a clinically significant abnormal pulmonary function test via spirometry [assessment by PI or delegate]
15. Has a COHb greater than 3%, or MetHb greater than 2% [measured by venous blood sample co-oximetry]

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, non-smoking volunteers ages 18-50 years who meet inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Accuracy root mean square | rSO2 and fSO2 data are recorded every 5-minutes during the procedure
  Accuracy root mean square is the square-root of the average squared distances between regional oxygen saturation (rSO2) as measured by INVOS and and field saturation (fSO2) as measured by blood sampling

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No